CLINICAL TRIAL: NCT00251771
Title: Catheter-directed Venous Thrombolysis in Acute Iliofemoral Vein Thrombosis, an Open Randomized, Controlled, Clinical Trial
Brief Title: Catheter-Directed Venous Thrombolysis in Acute Iliofemoral Vein Thrombosis
Acronym: CaVenT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.2005.650; EUDRACT No.2005-004486-42
Record Dates: First submitted 2005-11-09; First posted 2005-11-10 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2014-11

CONDITIONS: Deep Vein Thrombosis
Keywords: Thrombolytic therapy; Postphlebitic syndrome; Venous thrombosis
MeSH Terms: conditions — Venous Thrombosis; Postphlebitic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental)
  Interventions: Procedure: catheter-directed venous thrombolysis
- II (No Intervention)

INTERVENTIONS:
Procedure: catheter-directed venous thrombolysis — catheter-directed continuous intravenous infusion of alteplase 0.01mg/kg/h and low-dose heparin. Max dose 20mg/24 h and up to 96 hrs.
  Arms: I

SUMMARY:
Deep vein thrombosis (DVT) is a severe disease, and conventional treatment with low molecular weight heparin (LMWH) and warfarin is associated with some degree of long-term sequelae, i.e. post-thrombotic syndrome (PTS). Catheter-directed thrombolytic (CDT) therapy has been introduced worldwide the last two decades. Reports have suggested a beneficial effect of this costly treatment, but there are no randomized clinical trials documenting its short- and long-term efficacy and safety. This multi-center study will randomize patients with acute iliofemoral vein thrombosis to either conventional treatment or CDT in addition to conventional treatment. Main outcome parameters are patency rates at 6 months and prevalence of PTS at 24 months. The main short-term hypothesis is that CDT of first-time acute DVT will increase patency of the affected segments after 6 months from <50% to >80%. The main long-term hypothesis is that CDT will improve long-term functional outcome, i.e. risk of PTS after 2 years from >25% to <10%.

ELIGIBILITY:
Inclusion Criteria:

* Onset of symptoms <21 days
* Objectively verified DVT of the femoral or common iliac veins or the combined iliofemoral segment
* Informed consent

Exclusion Criteria:

* Anticoagulant therapy prior to trial entry >7 days
* Contraindications to thrombolytic therapy
* Indications for thrombolytic therapy, i.e. phlegmasia coerulea dolens or vena cava thrombosis
* Severe anemia, hemoglobin (hgb)<8 g/dl
* Thrombocytopenia, platelets <80x10^9/l
* Severe renal failure, creatinine clearance <30ml/min
* Severe hypertension, systolic (syst) blood pressure (BP)>160 mmHg or diastolic (diast) BP >100 mmHg pregnancy
* Less than 14 days post-surgery or post-trauma
* History of subarachnoidal or intracerebral bleeding
* Disease with life expectancy <24 months
* Drug abuse or mental disease that may interfere with treatment and follow-up
* Former ipsilateral proximal DVT
* Chemotherapy or advanced malignant disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2006-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Patency after 6 months | 6 months
Post-thrombotic syndrome after 2 years (yrs) | 2 years

SECONDARY OUTCOMES:
Frequency of clinically relevant bleeding complications | 1 year
Effects on quality of life | 2 and 5 years
Cost-effectiveness of treatment | 2 years
Procedural success of CDT | 1 week
Patency at 2 years | 2 years
PTS at 6, 12, 36, 48 and 60 months | 6, 12, 36, 48 and 60 months
Relation between PTS and patency | 2 years
Prevalence of vein anomalies | 6 months
Prevalence of underlying thrombophilia | 1 year
Frequency of recurrent venous thrombotic events (VTE) | 0.5, 2 and 5 years
Markers of importance for recurrent thrombosis | 0.5, 2 and 5 years
Markers of importance for successful thrombolysis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Per Morten Sandset, MD, Study Director — Ullevaal University Hospital
Locations (1):
- Ullevaal University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Enden T, Klow NE, Sandset PM. [Catheter-directed thrombolysis in acute deep venous thrombosis]. Tidsskr Nor Laegeforen. 2006 Jun 22;126(13):1765. No abstract available. Norwegian. PMID 16794675
- [Background] Enden T, Sandvik L, Klow NE, Hafsahl G, Holme PA, Holmen LO, Ghanima W, Njaastad AM, Sandbaek G, Slagsvold CE, Sandset PM. Catheter-directed Venous Thrombolysis in acute iliofemoral vein thrombosis--the CaVenT study: rationale and design of a multicenter, randomized, controlled, clinical trial (NCT00251771). Am Heart J. 2007 Nov;154(5):808-14. doi: 10.1016/j.ahj.2007.07.010. Epub 2007 Sep 6. PMID 17967583
- [Background] Enden T, Garratt AM, Klow NE, Sandset PM. Assessing burden of illness following acute deep vein thrombosis: data quality, reliability and validity of the Norwegian version of VEINES-QOL/Sym, a disease-specific questionnaire. Scand J Caring Sci. 2009 Jun;23(2):369-74. doi: 10.1111/j.1471-6712.2008.00618.x. Epub 2008 Nov 12. PMID 19068041
- [Background] Enden T, Sandset PM, Klow NE. Evidence-based practice for patients with severe venous thrombosis. Tidsskr Nor Laegeforen. 2012 May 29;132(10):1215-6. doi: 10.4045/tidsskr.12.0474. No abstract available. English, Norwegian. PMID 22669381
- [Result] Enden T, Klow NE, Sandvik L, Slagsvold CE, Ghanima W, Hafsahl G, Holme PA, Holmen LO, Njaastad AM, Sandbaek G, Sandset PM; CaVenT study group. Catheter-directed thrombolysis vs. anticoagulant therapy alone in deep vein thrombosis: results of an open randomized, controlled trial reporting on short-term patency. J Thromb Haemost. 2009 Aug;7(8):1268-75. doi: 10.1111/j.1538-7836.2009.03464.x. Epub 2009 Apr 30. PMID 19422443
- [Result] Enden T, Haig Y, Klow NE, Slagsvold CE, Sandvik L, Ghanima W, Hafsahl G, Holme PA, Holmen LO, Njaastad AM, Sandbaek G, Sandset PM; CaVenT Study Group. Long-term outcome after additional catheter-directed thrombolysis versus standard treatment for acute iliofemoral deep vein thrombosis (the CaVenT study): a randomised controlled trial. Lancet. 2012 Jan 7;379(9810):31-8. doi: 10.1016/S0140-6736(11)61753-4. Epub 2011 Dec 13. PMID 22172244
- [Result] Haig Y, Enden T, Slagsvold CE, Sandvik L, Sandset PM, Klow NE. Determinants of early and long-term efficacy of catheter-directed thrombolysis in proximal deep vein thrombosis. J Vasc Interv Radiol. 2013 Jan;24(1):17-24; quiz 26. doi: 10.1016/j.jvir.2012.09.023. Epub 2012 Nov 22. PMID 23176966
- [Result] Enden T, Resch S, White C, Wik HS, Klow NE, Sandset PM. Cost-effectiveness of additional catheter-directed thrombolysis for deep vein thrombosis. J Thromb Haemost. 2013 Jun;11(6):1032-42. doi: 10.1111/jth.12184. PMID 23452204
- [Result] Enden T, Wik HS, Kvam AK, Haig Y, Klow NE, Sandset PM. Health-related quality of life after catheter-directed thrombolysis for deep vein thrombosis: secondary outcomes of the randomised, non-blinded, parallel-group CaVenT study. BMJ Open. 2013 Aug 29;3(8):e002984. doi: 10.1136/bmjopen-2013-002984. PMID 23988361
- [Result] Enden T, Klow NE, Sandset PM. Symptom burden and job absenteeism after treatment with additional catheter-directed thrombolysis for deep vein thrombosis. Patient Relat Outcome Meas. 2013 Sep 16;4:55-9. doi: 10.2147/PROM.S47233. eCollection 2013. PMID 24082798
- [Derived] Flumignan RL, Nakano LC, Flumignan CD, Baptista-Silva JC. Angioplasty or stenting for deep venous thrombosis. Cochrane Database Syst Rev. 2025 Feb 19;2(2):CD011468. doi: 10.1002/14651858.CD011468.pub2. PMID 39968829
- [Derived] Broderick C, Watson L, Armon MP. Thrombolytic strategies versus standard anticoagulation for acute deep vein thrombosis of the lower limb. Cochrane Database Syst Rev. 2021 Jan 19;1(1):CD002783. doi: 10.1002/14651858.CD002783.pub5. PMID 33464575
- [Derived] Haig Y, Enden T, Grotta O, Klow NE, Slagsvold CE, Ghanima W, Sandvik L, Hafsahl G, Holme PA, Holmen LO, Njaaastad AM, Sandbaek G, Sandset PM; CaVenT Study Group. Post-thrombotic syndrome after catheter-directed thrombolysis for deep vein thrombosis (CaVenT): 5-year follow-up results of an open-label, randomised controlled trial. Lancet Haematol. 2016 Feb;3(2):e64-71. doi: 10.1016/S2352-3026(15)00248-3. Epub 2016 Jan 6. PMID 26853645
- See also: Protocol Reviews in the Lancet.com — http://www.thelancet.com/journals/lancet/misc/protocol/07PRT-295